CLINICAL TRIAL: NCT04214717
Title: Study of Dendritic Cell-activated Cytokine-induced Killer Cell Combined With Chemotherapy for Advanced Solid Tumor
Brief Title: Study of DC-CIK Combined With Chemotherapy for Advanced Solid Tumor
Acronym: DC-CIK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yantai Yuhuangding Hospital (Other)
Responsible Party: Principal Investigator, Peiwen Lian, Principle Investigator, Yantai Yuhuangding Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-008
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of DC-CIK with chemotherapy group (Experimental): Patients will receive DC-CIK treatments combined with Chemotherapy .
  Interventions: Combination Product: DC-CIK combined with Chemotherapy
- Chemotherapy group (Active Comparator): Patients will only receive Chemotherapy.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Combination Product: DC-CIK combined with Chemotherapy — Patients will receive 4 cycles of DC-CIK treatments combined with Chemotherapy within 8 months.
  Arms: Combination of DC-CIK with chemotherapy group
Drug: Chemotherapy — Patients will only receive Chemotherapy.
  Arms: Chemotherapy group

SUMMARY:
Combinations of Dendritic cell-activated cytokine-induced killer cell (DC-CIK) With chemotherapy treatment may enhance the immune response and stop cancer cells from growing.

DETAILED DESCRIPTION:
Patients in group A will receive 4 cycles of DC-CIK treatments within 8 months. Patients in group B will have no immunotherapy. Chemotherapy are available in both groups.The investigators want to evaluate the efficacy of combination of DC-CIK with chemotherapy in patients with treatment-refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with treatment-refractory advanced solid cancer can not accept operation;
2. Age 10 to 90 years;
3. Eastern Cooperative Oncology Group (ECOG) score ≤ 2 points;
4. Estimate survival > 3 months;
5. Blood White Blood Cell(WBC)≥ 4×109/L, Hb ≥ 100g/L, Platelet Count (PLT)≥ 80×109/L; Alanine amino transferase (ALT) and aspartate amino transferase (AST)≤ 2 times of normal upper value; Serum Cr ≤ 2 normal upper value;
6. Without any other malignant disease;
7. With more than one scalable lesions;
8. Patients Voluntary attempt, and informed consent;
9. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.

Exclusion Criteria:

1. Patients who do not conform to the inclusion criteria;
2. Patients with uncontrolled infection; underlying disease that was severe or life-threatening (such as uncontrolled brain metastasis );
3. Patients who were pregnant or lactating;
4. ECOG perform status ≥ 2;4.
5. Other situations that the researchers considered unsuitable for this study (such as mental illness, drug abuse, etc.)

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rates (DCR) | 1 year
  Disease Control Rates (Complete Remission + Partial Remission + Stable Disease), according to solid tumor response evaluation standard (Response evaluation criteria in solid tumors, RECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Peiwen Lian, PhD, Study Director — Yantai Yuhuangding Hospital
Locations (1):
- Yantai Yuhuangding Hospital, Yantai, Shandong, China

IPD SHARING:
Plan to Share IPD: No